CLINICAL TRIAL: NCT05351658
Title: Safety and Effectiveness of the External Fastening System for Temporary Active Fixation Pacemakers (TEMPACE)
Acronym: TEMPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ICU Medical Technologies S.L. (Industry)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TEMPACE
Record Dates: First submitted 2022-03-28; First posted 2022-04-28 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Arrythmia; Bradycardia
Keywords: Pacemaker; Cardiac pacing; Bradycardia; Arrhythmia; Treatment outcome
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Intervention Model Description: The study will be carried out in an Arrhythmia Unit or Intensive Care Unit. Patients who need urgent temporary cardiac pacing due to bradycardia, or elective pacing to prevent heart rhythm disturbances during high-risk arrhythmia interventions, such as transcatheter aortic valve implantation (TAVR), alcoholic septal ablations, etc., will be included. After the temporary pacemaker implantation with active fixation electrode in a correct way, the KronoSafe® external pacemaker fixation system will be placed. The correct functioning of the system (R wave detection, lead impedance and right ventricle threshold) will be checked at 24 hours and every other day until the end of cardiac stimulation. During temporary pacing, associated complications are going to be recorded: lead displacement, capture or sensing failure, generator or lead detachment, and cardiac perforation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporary Cardiac Pacing with Active-Fixation Leads (Experimental)
  Interventions: Device: KronoSafe® System

INTERVENTIONS:
Device: KronoSafe® System — All patients included in the study will have a temporary pacemaker with active fixation leads, held by the KronoSafe® fixation system.

SUMMARY:
Temporary cardiac pacing with active-fixation leads (TPAFL) using a reusable permanent pacemaker generator has been shown to be safer than lead systems without fixation. However, TPAFL requires the off-label (non-certificated) use of Pacemaker leads and generators. It is designed a fastening system to ensure the safety and efficacy of the procedure: the KronoSafe System®. The aim of this study is to demonstrate the safety and effectiveness of the KronoSafe System® for temporary pacing in a series of patients receiving TPAFL.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Need for temporary cardiac stimulation
* Temporary active fixation pacemaker implantation through left or right jugular access.
* Signature of informed consent
* Correct functioning of the electrode after the implantation: sensing of the R wave above 5 millivolts. Ventricular pacing threshold below 1 volt. Electrode impedance between 400-1200 Ohm.
* Pacemaker programming with stimulation output at 5 volts intensity and 1 millisecond pulse duration.
* Placement of the KronoSafe® fastening system after electrode implantation.

Exclusion Criteria:

* Complication during the procedure: pneumothorax, hematoma at the puncture site, cardiac perforation, accidental arterial puncture or other that, in the investigator's opinion, poses an added risk of pacemaker dysfunction.
* Need to transfer the patient to another center with loss of follow-up.
* Absence of surveillance through continuous electrocardiographic monitoring with detection of arrhythmic events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Ventricular R wave detection | Immediately after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Lead impedance detection | Immediately after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Right ventricle threshold detection | Immediately after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Ventricular R wave detection | 24 hours after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 3 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 5 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 7 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 9 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 11 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 13 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 15 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 17 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 19 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 21 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 23 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 25 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 27 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | day 29 after the procedure of lead implantation
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Ventricular R wave detection | Immediately before the procedure of lead removal
  Ventricular R wave, measured in millivolts with pacemaker generator programmer
Lead impedance detection | 24 hours after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 3 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 5 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 7 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 9 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 11 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 13 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 15 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 17 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 19 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 21 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 23 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 25 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 27 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | day 29 after the procedure of lead implantation
  Lead impedance, measured in ohms with pacemaker generator programmer
Lead impedance detection | Immediately before the procedure of lead removal
  Lead impedance, measured in ohms with pacemaker generator programmer
Right ventricle threshold detection | 24 hours after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 3 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 5 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 7 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 9 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 11 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 13 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 15 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 17 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 19 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 21 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 23 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 25 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 27 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | day 29 after the procedure of lead implantation
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Right ventricle threshold detection | Immediately before the procedure of lead removal
  Right ventricle threshold, measured in volts with pacemaker generator programmer
Lead displacement detection | Immediately before the procedure of lead removal
  Visual observation of 2 cm electrode displacement through vein acces by clinical examination
Capture failure detection | Immediately before the procedure of lead removal
  Right ventricle threshold above 5 volts during 1 millisecond, measured with pacemaker generator programmer.
Sensing failure detection | Immediately before the procedure of lead removal
  Ventricular R wave below 1 volt, measured with pacemaker generator programmer
Lead insulation breakdown detection | Immediately before the procedure of lead removal
  Visual observation of lead insulation breakdown by clinical examination
Generator detachment detection | Immediately before the procedure of lead removal
  Visual observation of generator detachment by clinical examination. removal of the generator from the casing.
Cardiac peroration detection | Immediately before the procedure of lead removal
  New pericardial effusion detected by Echocardiography with signs of cardiac tamponade: respiratory variation of transmitral filling flow greater than 25%

SECONDARY OUTCOMES:
Detection of Bacteremia | Immediately after the procedure of lead removal
  Isolation of the same bacteria in the pacemaker lead and 2 blood cultures from the patient
Detection of Agitation | Immediately after the procedure of lead removal
  Record of antipsychotic and anxiolytic treatment of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Raimundo Vicente, MD, Principal Investigator — Intensive Care Physician at Dr. Balmis University Hospital (Alicante)
Locations (2):
- Spain (2):
  - Hospital General Universitario de Alicante Dr.Balmis, Alicante
  - Hospital Universitari Vall D'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vicente-Miralles R, Martin-Langerwerf DA, Nunez-Martinez JM, Marco-Juan A, Sangio-Ferreyros AD, Davila-Arias A, Montes-Jacobo L, Barrios V, Palazon-Bru A, Gil-Guillen VF, Bertomeu-Gonzalez V. A new fastening system for temporary pacing with active-fixation leads: effectiveness and safety. Eur Heart J Acute Cardiovasc Care. 2022 Mar 16;11(3):224-229. doi: 10.1093/ehjacc/zuab119. PMID 34918044
- [Result] Zei PC, Eckart RE, Epstein LM. Modified temporary cardiac pacing using transvenous active fixation leads and external re-sterilized pulse generators. J Am Coll Cardiol. 2006 Apr 4;47(7):1487-9. doi: 10.1016/j.jacc.2006.01.006. Epub 2006 Mar 15. No abstract available. PMID 16580542
- [Result] Kawata H, Pretorius V, Phan H, Mulpuru S, Gadiyaram V, Patel J, Steltzner D, Krummen D, Feld G, Birgersdotter-Green U. Utility and safety of temporary pacing using active fixation leads and externalized re-usable permanent pacemakers after lead extraction. Europace. 2013 Sep;15(9):1287-91. doi: 10.1093/europace/eut045. Epub 2013 Mar 12. PMID 23482613
- [Result] Betts TR. Regional survey of temporary transvenous pacing procedures and complications. Postgrad Med J. 2003 Aug;79(934):463-5. doi: 10.1136/pmj.79.934.463. PMID 12954959
- [Derived] Vicente-Miralles R, Rivas-Gandara N, Jordan Marchite P, Adelino R, Carmona MA, Diaz Barranco M, Ibanez Criado AA, Ruiz Nodar JM, Ajo Ferrer M, Garcia-Fernandez A, Bertomeu-Gonzalez V, Martinez Martinez JG. A Novel Device for Temporary Cardiac Stimulation Using Permanent Pacemaker Generators and Active-Fixation Leads: The TEMPACE Multi-Center Prospective Study. Eur Heart J Acute Cardiovasc Care. 2025 Aug 28:zuaf111. doi: 10.1093/ehjacc/zuaf111. Online ahead of print. PMID 40875828